CLINICAL TRIAL: NCT02111993
Title: Evaluating Myocardial Injury During ICD Implantation Using the Upper Limit of Vulnerability (ULV) Method vs. Standard Defibrillation Threshold Testing
Brief Title: Evaluating Myocardial Injury for Defibrillation Threshold Testing Methods for ICD Implantation
Acronym: ULV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Ulrika Birgersdotter-Green, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 110647
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Cardiomyopathy; Heart Failure; Cardiac Arrhythmia
Keywords: Defibrillation testing; Upper Limit of Vulnerability; ULV; DFT; ICD; implantable cardioverter defibrillator; cardiomyopathy; cardiac arrhythmia; cardiac device testing
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Defibrillation Testing (Active Comparator): Standard Defibrillation Threshold Testing is a procedure in which a low energy shock will be delivered to the heart to induce ventricular fibrillation (VF) followed by a rescue shock to restore sinus rhythm. Process is repeated after 5 minutes.
  Interventions: Device: Standard Defibrillation Testing
- Upper Limit of VulnerabilityTesting (Active Comparator): Upper Limit of Vulnerability Testing is a procedure in which four 18J shocks will be delivered at specified intervals. If VF is induced, then a 25 J rescue shock will be delivered.
  Interventions: Device: Upper Limit of Vulnerability Testing

INTERVENTIONS:
Device: Standard Defibrillation Testing — Once the ICD is implanted, Standard Defibrillation Threshold (DFT) testing will begin. A low energy shock will be delivered to the heart at the peak of the T wave to induce ventricular fibrillation (VF). Once VF is induced, a rescue shock of 25J will be delivered to restore sinus rhythm. This process will be repeated once more after 5 minutes.
  Other Names: ICD implantation
  Arms: Standard Defibrillation Testing
Device: Upper Limit of Vulnerability Testing — Once the ICD is implanted, Upper Limit of Vulnerability (ULV) testing will commence. An 18 J shock will be delivered will at different points from the t-wave. If VF is not induced with any of these shocks, then the ULV will be considered to be 18J. If VF is induced, then a 25 J rescue shock will be delivered.
  Other Names: ICD implantation
  Arms: Upper Limit of VulnerabilityTesting

SUMMARY:
The objective of this study is to evaluate myocardial injury, if any, as quantified by cardiac markers (Troponin-T) in defibrillation threshold (DFT) testing during implantation of implantable cardioverter defibrillators (ICDs) using the upper limit of vulnerability (ULV) method vs. standard defibrillation threshold method.

DETAILED DESCRIPTION:
This is a prospective, randomized (1:1 DFT vs ULV testing), controlled clinical research trial. Patients undergoing ICD implant or device change out will be candidates for this study. Medical records for these patients will be screened prior to enrollment to ensure eligibility for the study. Each patient who is a candidate and who agrees to participate in the study will undergo the standard of care pre-procedure evaluation including a complete medical history evaluation, a complete physical examination and routine laboratory testing including chemistry panel, hematology panel, coagulation panel, a 12-lead electrocardiogram, and a urine pregnancy test (all females of child-bearing age). A candidate patient will be randomly assigned to either the standard DFT testing method group or the ULV testing method group.

For the standard DFT testing group, per routine standard of care, the patient will be admitted to the hospital. The study requires a pre-procedure blood test of 3 ml for Troponin-T (TnT) which will be drawn prior to any DFT testing. The blood sample will be sent to the University of California, San Diego (UCSD) central laboratory for processing. The patient will then undergo the scheduled ICD implant procedure in a standard fashion. The standard defibrillation threshold testing will be performed using a low energy shock delivered on T-wave to induce ventricular fibrillation (VF). If VF is induced, the first shock is 25 Joules (J). If success, we will wait 5 minutes and repeat the process. If the 2nd shock yields success, the DFT testing is complete and a 10J safety margin achieved (device shock energy is set at 35J or as clinically indicated determined by treating Cardiac Electrophysiologist). A back-up external defibrillator will always be immediately available in case transvenous shocks fail. Blood pressure will be monitored before and immediately after each shock. After 4 hours, 8 hours and 16 hours post DFT testing, blood samples (3 ml for Troponin-T) will be drawn and sent to the UCSD central laboratory for processing.

For the ULV testing group, per routine standard of care, the patient will be admitted to the hospital. The study requires a pre-procedure blood test (3 ml for Troponin-T.) which will be drawn prior to any ULV testing. The blood sample will be sent to the UCSD central laboratory for processing. The patient will then undergo the scheduled ICD implant procedure as is standard clinical care. The ULV testing is performed as follows: for single coil device, a 18J shock will be delivered at 0msec, +20 msec, -20msec and -40msec measured from the peak of the T-wave; for dual coil device, a 18J shock will be delivered at 0msec, -20msec, +20msec, and +40msec measured from the peak of the T-wave. If VF is not induced with any of the above mentioned shocks, the ULV will be considered as 18J and the ICD will be implanted with the first shock strength set at 30 joules or as clinically indicated determined by treating Cardiac Electrophysiologist. If VF is induced, a 25J rescue shock will be delivered as is standard and if successful, the device will be programmed to the maximum output of 35 joules or as clinically indicated determined by treating Cardiac Electrophysiologist. Blood pressure will be monitored before and immediately after each shock. After 4 hours, 8 hours and 16 hours post ULV testing, blood samples (3 ml for Troponin-T) will be drawn and sent to the UCSD central laboratory for processing.

Other than the blood tests for Troponin-T, there is no change in routine post-operative management. Patients will be followed every three months, as is standard management for patients with ICDs.

The TnT blood draws at 4-hour, 8-hour and 16-hour post implantation will not require longer hospital stay than is standard for patients undergoing ICD implantation. The results of Troponin-T measurement for the study patients will be reviewed by the cardiac electrophysiology (EP) research staff. If myocardial injury is noted (any TnT value >0.1 as per current assay at the UCSD laboratory), the patient will be monitored as is deemed clinically necessary by treating Cardiac Electrophysiologist, including possible repeat TnT measurements for evaluation of myocardial infarction. We will follow standard of care for management of myocardial injury as recommended by the American Heart Association and the American College of Cardiology. Elevated TnT measurements may delay hospitalization, if determined to be clinically necessary. If the repeat TnT measurement is <0.1, then myocardial injury is most unlikely and the positive TnT value is likely due to DFT shocks.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible to receive an ICD implant or change out.
* Patients with a single or dual coil right ventricle (RV) defibrillation lead located in the RV apex.
* Patients greater than 18 years of age.
* Patients willing and able to give informed consent.
* Patients who have insurance which may cover additional hospital stay if myocardial injury resulted from testing

Exclusion Criteria:

* Patients with medical conditions that would limit study participation.
* Patients that are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Birgersdotter-Green, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Sulpizio Cardiovascular Center, La Jolla, California, United States

REFERENCES:
- [Background] Swerdlow CD, Shehata M, Chen PS. Using the upper limit of vulnerability to assess defibrillation efficacy at implantation of ICDs. Pacing Clin Electrophysiol. 2007 Feb;30(2):258-70. doi: 10.1111/j.1540-8159.2007.00659.x. PMID 17338725
- [Background] Day JD, Doshi RN, Belott P, Birgersdotter-Green U, Behboodikhah M, Ott P, Glatter KA, Tobias S, Frumin H, Lee BK, Merillat J, Wiener I, Wang S, Grogin H, Chun S, Patrawalla R, Crandall B, Osborn JS, Weiss JP, Lappe DL, Neuman S. Inductionless or limited shock testing is possible in most patients with implantable cardioverter- defibrillators/cardiac resynchronization therapy defibrillators: results of the multicenter ASSURE Study (Arrhythmia Single Shock Defibrillation Threshold Testing Versus Upper Limit of Vulnerability: Risk Reduction Evaluation With Implantable Cardioverter-Defibrillator Implantations). Circulation. 2007 May 8;115(18):2382-9. doi: 10.1161/CIRCULATIONAHA.106.663112. Epub 2007 Apr 30. PMID 17470697
- [Background] Chen PS, Shibata N, Dixon EG, Martin RO, Ideker RE. Comparison of the defibrillation threshold and the upper limit of ventricular vulnerability. Circulation. 1986 May;73(5):1022-8. doi: 10.1161/01.cir.73.5.1022. PMID 3698224
- [Background] Chen PS, Feld GK, Kriett JM, Mower MM, Tarazi RY, Fleck RP, Swerdlow CD, Gang ES, Kass RM. Relation between upper limit of vulnerability and defibrillation threshold in humans. Circulation. 1993 Jul;88(1):186-92. doi: 10.1161/01.cir.88.1.186. PMID 8319332
- [Background] Hwang C, Swerdlow CD, Kass RM, Gang ES, Mandel WJ, Peter CT, Chen PS. Upper limit of vulnerability reliably predicts the defibrillation threshold in humans. Circulation. 1994 Nov;90(5):2308-14. doi: 10.1161/01.cir.90.5.2308. PMID 7955188
- [Background] Martin DJ, Chen PS, Hwang C, Gang ES, Mandel WJ, Peter CT, Swerdlow CD. Upper limit of vulnerability predicts chronic defibrillation threshold for transvenous implantable defibrillators. J Cardiovasc Electrophysiol. 1997 Mar;8(3):241-8. doi: 10.1111/j.1540-8167.1997.tb00786.x. PMID 9083873
- [Background] Birgersdotter-Green U, Undesser K, Fujimura O, Feld GK, Kass RM, Mandel WJ, Peter CT, Chen PS. Correlation of acute and chronic defibrillation threshold with upper limit of vulnerability determined in normal sinus rhythm. J Interv Card Electrophysiol. 1999 Jul;3(2):155-61. doi: 10.1023/a:1009825731592. PMID 10387143
- [Background] Swerdlow CD, Davie S, Ahern T, Chen PS. Comparative reproducibility of defibrillation threshold and upper limit of vulnerability. Pacing Clin Electrophysiol. 1996 Dec;19(12 Pt 1):2103-11. doi: 10.1111/j.1540-8159.1996.tb03285.x. PMID 8994950
- [Background] Swerdlow CD, Ahern T, Kass RM, Davie S, Mandel WJ, Chen PS. Upper limit of vulnerability is a good estimator of shock strength associated with 90% probability of successful defibrillation in humans with transvenous implantable cardioverter-defibrillators. J Am Coll Cardiol. 1996 Apr;27(5):1112-8. doi: 10.1016/0735-1097(95)00603-6. PMID 8609329
- [Background] Swerdlow CD. Implantation of cardioverter defibrillators without induction of ventricular fibrillation. Circulation. 2001 May 1;103(17):2159-64. doi: 10.1161/01.cir.103.17.2159. PMID 11331256
- [Background] Green UB, Garg A, Al-Kandari F, Ungab G, Tone L, Feld GK. Successful implantation of cardiac defibrillators without induction of ventricular fibrillation using upper limit of vulnerability testing. J Interv Card Electrophysiol. 2003 Feb;8(1):71-5. doi: 10.1023/a:1022304417889. PMID 12652181
- [Background] Swerdlow C, Shivkumar K, Zhang J. Determination of the upper limit of vulnerability using implantable cardioverter-defibrillator electrograms. Circulation. 2003 Jun 24;107(24):3028-33. doi: 10.1161/01.CIR.0000074220.19414.18. Epub 2003 Jun 16. PMID 12810611
- [Background] Shehata M, Belk P, Kremers M, Saba S, Cao J, Swerdlow CD. Automatic determination of timing intervals for upper limit of vulnerability using ICD electrograms. Pacing Clin Electrophysiol. 2008 Jun;31(6):691-700. doi: 10.1111/j.1540-8159.2008.01072.x. PMID 18507541

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 patients were consented and enrolled in this trial. 9 of which were withdrawn due to incomplete lab draws. 51 patients successfully completed study procedures and were included in the study data analysis.
Period: Overall Study
Arm/Group | Standard Defibrillation Testing | Upper Limit of VulnerabilityTesting
Started | 30 | 30
Completed | 25 | 26
Not Completed | 5 | 4
Not completed — Physician Decision | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Defibrillation Testing | Upper Limit of VulnerabilityTesting | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (16) | 63 (11) | 65 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 19 | 21 | 40
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (7.0) | 27.4 (4.6) | 27.8 (5.1)
History of Hypertension (HTN) [Number; unit: participants] | 16 | 12 | 28
Presence of Left Ventricular Hypertrophy (LVH) [Number; unit: participants] | 9 | 17 | 26
History of Ventricular Tachycardia (VT) [Number; unit: participants] | 8 | 10 | 18
History of Non-Ischemic Cardiomyopathy (NICM) [Number; unit: participants] | 2 | 6 | 8
History of Diabetes Mellitus (DM) [Number; unit: participants] | 5 | 6 | 11
History of Coronary Artery Bypass Graft (CABG) [Number; unit: participants] | 4 | 1 | 5
Secondary Prevention Implanted Cardiac Defibrillator (ICD) [Number; unit: participants] | 2 | 1 | 3
Anti-Arrhythmic Medication [Number; unit: participants] | 5 | 6 | 11
Beta-Blocker Medication [Number; unit: participants] | 15 | 19 | 34
Ejection Fraction (EF) (%) [Mean (Standard Deviation); unit: percentage] | 40 (17) | 34 (18) | 38 (17.6)
End Diastolic Volume (EDV) [Mean (Standard Deviation); unit: cm] | 5.4 (0.9) | 5.5 (1.1) | 5.45 (1.0)
Dual Coil ICD [Number; unit: participants] | 12 | 10 | 22
Single Coil ICD [Number; unit: participants] | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Damage
Description: Myocardial damage will be evaluated by cardiac troponin (cTNT) lab collection before and then after ULV or DFT testing at 4 hours, 8 hours, and 20 hours.
Time Frame: 20 hours (hr)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Standard Defibrillation Testing | Upper Limit of VulnerabilityTesting
Number analyzed (Participants) | 25 | 26
ng/mL
  Δ4 hr cTnT | 0.001 (0.023) | 0.011 (0.066)
  Δ8 hr cTnT | 0.002 (0.030) | 0.012 (0.072)
  Δ20 hr cTnT | 0.002 (0.032) | 0.001 (0.048)
Statistical Analysis 1: Comparison: Standard Defibrillation Testing vs Upper Limit of VulnerabilityTesting; Test type: Superiority or Other; p = 0.02, t-test, 2 sided — This p-value correlates to Δ4 hr cTnT
Statistical Analysis 2: Comparison: Standard Defibrillation Testing vs Upper Limit of VulnerabilityTesting; Test type: Superiority or Other; p = 0.03, t-test, 2 sided — This p-value correlates to Δ8 hr cTnT
Statistical Analysis 3: Comparison: Standard Defibrillation Testing vs Upper Limit of VulnerabilityTesting; Test type: Superiority or Other; p = 0.16, t-test, 2 sided — This p-value correlates to Δ20 hr cTnT

2. Secondary Outcome: Defibrillation Testings (DFT) vs. Upper Limit of Vulnerability (ULV) (VF Induced)
Description: the DFT group cardiac troponin (cTNT) values were compared to the subjects within the ULV group that required VF induction.
Time Frame: 20 hours (hr)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Upper Limit of VulnerabilityTesting (VF Induced): Upper Limit of Vulnerability Testing is a procedure in which four 18J shocks will be delivered at specified intervals. If VF is induced, then a 25 J rescue shock will be delivered.
  Upper Limit of Vulnerability Testing: Once the ICD is implanted, Upper Limit of Vulnerability (ULV) testing will commence. An 18 J shock will be delivered will at different points from the t-wave. VF was induced in a subset of the ULV patients, and a 25 J rescue shock was delivered.
Arm/Group | Standard Defibrillation Testing | Upper Limit of VulnerabilityTesting (VF Induced)
Number analyzed (Participants) | 25 | 11
ng/mL
  Δ4 hr cTnT | 0.001 (0.023) | 0.075 (0.086)
  Δ8 hr cTnT | 0.002 (0.030) | 0.078 (0.093)
  Δ20 hr cTnT | 0.002 (0.032) | 0.042 (0.057)
Statistical Analysis 1: Comparison: Standard Defibrillation Testing vs Upper Limit of VulnerabilityTesting (VF Induced); Test type: Superiority or Other; p = 0.04, t-test, 2 sided — This p-value correlates to Δ4 hr cTnT
Statistical Analysis 2: Comparison: Standard Defibrillation Testing vs Upper Limit of VulnerabilityTesting (VF Induced); Test type: Superiority or Other; p = 0.06, t-test, 2 sided — This p-value correlates to Δ8 hr cTnT
Statistical Analysis 3: Comparison: Standard Defibrillation Testing vs Upper Limit of VulnerabilityTesting (VF Induced); Test type: Superiority or Other; p = 0.16, t-test, 2 sided — This p-value correlates to Δ20 hr cTnT

3. Secondary Outcome: Defibrillation Testing (DFT) Versus Upper Limit of Vulnerability (ULV) (Non-induced)
Description: The DFT group was compared to the ULV subgroup that did not require ventricular fibrillation (VF) induction. Cardiac troponin (cTNT) levels were analyzed.
Time Frame: 20 hours (hr)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Upper Limit of VulnerabilityTesting (No VF Induction): Upper Limit of Vulnerability Testing is a procedure in which four 18J shocks will be delivered at specified intervals. If VF is induced, then a 25 J rescue shock will be delivered.
  Upper Limit of Vulnerability Testing: Once the ICD is implanted, Upper Limit of Vulnerability (ULV) testing will commence. An 18 J shock will be delivered will at different points from the t-wave. VF was not induced in this subgroup with any of these shocks, and the ULV was considered to be 18J.
Arm/Group | Standard Defibrillation Testing | Upper Limit of VulnerabilityTesting (No VF Induction)
Number analyzed (Participants) | 25 | 14
ng/mL
  Δ4 hr cTnT | 0.001 (0.023) | 0.031 (0.031)
  Δ8 hr cTnT | 0.002 (0.030) | 0.038 (0.038)
  Δ20 hr cTnT | 0.002 (0.032) | 0.031 (0.031)
Statistical Analysis 1: Comparison: Standard Defibrillation Testing vs Upper Limit of VulnerabilityTesting (No VF Induction); Test type: Superiority or Other; p = 0.17, t-test, 2 sided — This p-value correlates to Δ4 hr cTnT
Statistical Analysis 2: Comparison: Standard Defibrillation Testing vs Upper Limit of VulnerabilityTesting (No VF Induction); Test type: Superiority or Other; p = 0.19, t-test, 2 sided — This p-value correlates to Δ8 hr cTnT
Statistical Analysis 3: Comparison: Standard Defibrillation Testing vs Upper Limit of VulnerabilityTesting (No VF Induction); Test type: Superiority or Other; p = 0.38, t-test, 2 sided — This p-value correlates to Δ20 hr cTnT

ADVERSE EVENTS:
Arm/Group | Standard Defibrillation Testing | Upper Limit of VulnerabilityTesting
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No